CLINICAL TRIAL: NCT05695612
Title: EVALUATION OF TWO DIFFERENT ATTACHMENT SYSTEMS IN MANDIBULAR OVERDENTURES RETAINED WITH TWO INCLINED IMPLANTS (A RANDOMIZED CONTROLLED CLINICAL TRIAL)
Brief Title: EVALUATION OF TWO DIFFERENT ATTACHMENT SYSTEMS IN MANDIBULAR OVERDENTURES RETAINED WITH TWO INCLINED IMPLANTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, haitham ahmed hassan ismail, Assistant Lecturer of Prosthodontics, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00010556-IORG0008839
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Inclined Implants

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novaloc Attachment (Experimental)
  Interventions: Other: Novaloc Attachment
- Locator attachment (Active Comparator)
  Interventions: Other: Locator Attachment

INTERVENTIONS:
Other: Novaloc Attachment — Each patient will receive two inclined implants placed in the mandibular canine region bilaterally using the flapless surgical technique. Patients will receive mandibular overdentures with Novaloc attachments. The proper Novaloc abutments will be selected and screwed on the implants according to the prosthetic platform and the tissue height. The metal housings will be connected to the existing mandibular overdenture by pick-up technique.
  Arms: Novaloc Attachment
Other: Locator Attachment — Each patient will receive two inclined implants placed in the mandibular canine region bilaterally using the flapless surgical technique. Patients will receive mandibular overdentures with Locator attachments. The proper Locator abutments will be selected and screwed on the implants according to the prosthetic platform and the tissue height. The metal housings will be connected to the existing mandibular overdenture by pick-up technique.
  Arms: Locator attachment

SUMMARY:
The aim of the study is to evaluate clinically and radiographically the Novaloc and Locator attachment systems in mandibular overdentures retained with two inclined implants.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be completely edentulous.
* Patients should have enough bone for the placement of implants at least 3.5 mm in diameter and 10.0 mm in length.
* Patients should be co-operative and have adequate dexterity for placement and removal of the implant -retained overdenture.
* The inter-ridge space should be sufficient to place the endosseous implants and the superstructures

Exclusion Criteria:

* Patients with any systematic disease that could complicate the surgical phase or affect osseointegration as osteoporosis and uncontrolled diabetes mellitus.
* Patients with active oral infections.
* Patients with history of radiotherapy in head and neck region.
* Patients with poor oral hygiene.
* Patients with restricted mouth openings ≤ 40mm, functional limitations, or temporo-mandibular disorders.
* Heavy smokers (more than 10 cigarette / day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Peri-implant Probing Depth (PD) | up to 12 months
  The distance from the gingival margin till the point of least resistance will be measured using a graduated plastic autoclavable periodontal probe. The probe will be held parallel to the long axis of the implant and introduced with light force to the peri-implant sulcus. Measurements will be made at 6 sites around each implant; mesiobuccal, mid-buccal, disto-buccal, mesio-palatal, mid-palatal and disto-palatal. Probing depth of 1 mm or less will be recorded as 1 mm, and those exceeding 1 mm, but less than 2 mm, will be recorded as 2 mm, and so on. The mean for each implant will be calculated.
Modified Sulcus Bleeding Index (BI) | up to 12 months
  This will be measured using a graduated plastic autoclavable periodontal probe. The probe will be held parallel to the long axis of the implant and introduced with light force to the peri-implant sulcus. A score of 0-3 will be assigned to each labial and palatal surface of the implant then the average for each implant will be calculated according to the following criteria:
  Score 0: No bleeding when a periodontal probe is passed along the gingival margin adjacent to the implant.
  Score 1: Isolated bleeding spots visible. Score 2: Blood forms a confluent red line on margin. Score 3: Heavy or profuse bleeding
Modified gingival index | up to 12 months
  The peri-implant mucosal tissues will be assessed according to Lobene and Weatherford as follows:
  0: Absence of inflammation, normal gingiva.
  1. Mild inflammation, slight color change, little change in texture of any portion of, but not entire, marginal, or papillary gingival unit (localized).
  2. Mild inflammation, slight color change, little change in texture involving the entire or papillary gingival unit (generalized)..
  3. Moderate inflammation, redness, and edema.
  4. Severe inflammation, marked redness, edema, ulceration, and spontaneous bleeding It will be measured at 4 sites around each implant (mesially, distally, labially/ buccaly, lingually) then, the mean record will be calculated for each implant. Indices of the two implants will be added to each other, and then divided by 2 to get the mean modified gingival index for each case.
Alveolar bone level | up to 12 months
  The level of alveolar bone around each implant will be assessed using CBCT(3D Accuitomo 170, 90 kVp, 5 mA, 30.8 s, 0.08 mm isotropic voxel size, J Morita, Kyoto, Japan) and the field of view will be the lower anterior sextant. The vertical bone change (distance from the implant platform to the first bone-to-implant contact, in mm) around each implant will be assessed at the buccal, lingual, mesial and distal aspects then the mean will be calculated.
Implant stability | up to 12 months
  Magnetic Resonance Frequency Analyser will be used to measure the implant stability quotient (ISQ). The instrument measures the resonance frequency through the transducer attached to a implant fixture and display the result ISQ value on a scale of 1 to 100 with higher values indicating higher stability. The measurements will be made three times and the mean will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Haitham Ismail, MSc, Principal Investigator — Alexandria University; Ahmed Al-Shimy, PhD, Study Director — Alexandria University; Tarek S Abdelazim, PhD, Study Chair — Alexandria University; Kenda IH Hanno, PhD, Study Chair — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt